CLINICAL TRIAL: NCT02940834
Title: Sodium Imbalance in Traumatic Brain Injury Patients: Prevalence,Predictors and Prognostic Significance in a Tertiary Care Centre
Brief Title: Sodium Imbalance in Traumatic Brain Injury Patients: Prevalence, Predictors and Prognostic Significance in a Tertiary Care Centre
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, DR GANESH ADAIKKALAVAN M, DR, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: Na TBI
Record Dates: First submitted 2016-10-18; First posted 2016-10-21 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Sodium Imbalance in Traumatic Brain Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients with sodium imbalance
- patients without sodium imbalance

SUMMARY:
Observational study about prevalence, predictors of sodium imbalance and prognostic significance.

ELIGIBILITY:
Inclusion Criteria:

* adult and paediatric patients with isolated head injury

Exclusion Criteria:

* age more than 80 years, patient admitted after 24 hours of trauma, chronic kidney disease, chronic liver disease, associated chest trauma, abdominal trauma

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: adult and paediatric patients with isolated traumatic brain injury admitted in ICU in PGIMER
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
correlate prevalence of sodium imbalance with severity of traumatic brain injury by biochemistry lab reports | first 10 days after admission in icu or discharge whichever is earlier

SECONDARY OUTCOMES:
predisposing factors for development of sodium imbalance in traumatic brain injury patients by logistic regression analysis of data | first 10 days after admission in icu or discharge whichever is earlier
relationship between sodium imbalance and outcome in traumatic brain injury patients by assessing Glasgow outcome score telephonically | 1st and 3rd month after discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Medical Education and Research, Chandigarh, Chandigarh, India